CLINICAL TRIAL: NCT02465073
Title: The Clinical Efficacy of Next Science Wound Gel (NXTSC) in the Healing of Chronic Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southwest Regional Wound Care Center (Other)
Collaborators: Next Science TM (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 56-RW-027
Record Dates: First submitted 2014-12-19; First posted 2015-06-08 (Estimated); Results first posted 2016-01-18 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Wound Infection
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- NXTSC (Active Comparator): This group will receive the NXTSC gel only. The NXTSC wound gel and its active agents are applied on the wound bed. A synthetic microfiber dressing will be applied to the surface of the wound. Determine the effect on wound treatment outcomes using a novel antimicrobial wound gel for the treatment of infected wounds as the sole topical treatment of microbial infection at the wound site. ( NXTSC).
  Interventions: Device: NXTSC wound gel
- NXTSC plus SOC (Active Comparator): This group will receive the NXTSC wound gel plus Standard of Care. The NXTSC wound gel is applied to the wound bed. Local wound management will consist of diagnosing the wound biofilm and providing specific measures to suppress the wound biofilm to allow host healing. Determine the effect on wound treatment outcomes using a novel antimicrobial wound gel for the treatment of infected wounds when this gel is used in conjunction with the current standard of care infection controls to treat microbial infection at the wound site.( Next Science Wound Gel, plus standard of care).
  Interventions: Device: NXTSC wound gel plus Standard of Care
- SOC (Active Comparator): This group will receive Standard of Care only. The Standard of Care is based on wound management intervention to remove wound slough by frequent debridement. Moist interactive wound care with multiple strategies to suppress biofilm is instituted. Determine the effect on wound treatment outcomes using standard of care treatment
  Interventions: Device: Standard of Care Group

INTERVENTIONS:
Device: NXTSC wound gel — Subjects will receive NXTSC wound gel only.
  Other Names: NXTSC
  Arms: NXTSC
Device: NXTSC wound gel plus Standard of Care — Subjects will be randomized to the NXTSC wound gel plus Standard of Care of only.
  Other Names: NXTSC + SOC
  Arms: NXTSC plus SOC
Device: Standard of Care Group — Subjects will receive Standard of Care only.
  Other Names: SOC
  Arms: SOC

SUMMARY:
Determine the effect on wound treatment outcomes using a novel antimicrobial wound gel (NXTSC) for the treatment of infected wounds as the sole topical treatment of microbial infection at the wound site.

DETAILED DESCRIPTION:
1. Determine the effect on wound treatment outcomes using a novel antimicrobial wound gel (NXTSC) for the treatment of infected wounds as the sole topical treatment of microbial infection at the wound site.
2. Determine the effect on wound treatment outcomes using a novel antimicrobial wound gel for the treatment of infected wounds when this gel is used in conjunction with the current standard of care infection controls to treat microbial infection at the wound site.
3. Determine the effect on wound treatment outcomes using standard of care treatment. (SOC).

ELIGIBILITY:
Inclusion Criteria:

1. The subject must have a full-thickness chronic wound for greater than one month.
2. The subject must be at least 18 years of age.
3. The ulcer to be biopsied must be greater than 1 centimeter in area.
4. The subject must be able to give informed consent.

Exclusion Criteria:

1. Medical or emotional risk associated with the potential biopsy that outweighs the risk of not taking a biopsy as determined by the investigator.
2. Those patients that have significant contributions from other disease processes such as arterial disease (Ankle Brachial Index [ABI] less than .7, OR Transcutaneous Partial Oxygen Pressure [TCpO2 ] less than 20) will be considered to have mixed vascular disease producing their wound and will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randall D Wolcott, M.D., Principal Investigator — Southwest Regional Wound Care Center
Locations (1):
- Southwest Regional Wound Care Center, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- NXTSC: This group will receive the NXTSC gel only.
  NXTSC wound gel: Subjects will receive NXTSC wound gel only.
- NXTSC Plus SOC: This group will receive the NXTSC wound gel plus Standard of Care.
  NXTSC wound gel plus Standard of Care: Subjects will be randomized to the NXTSC wound gel plus Standard of Care of only.
- Standard of Care: This group will receive Standard of Care only.
  Standard of Care Group: Subjects will receive Standard of Care only.
Period: Overall Study
Arm/Group | NXTSC | NXTSC Plus SOC | Standard of Care
Started | 17 | 16 | 16
Completed | 15 | 15 | 15
Not Completed | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NXTSC | NXTSC Plus SOC | Standard of Care | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 13 | 12 | 34
  >=65 years | 6 | 2 | 3 | 11
Age, Continuous [Mean (Full Range); unit: years] | 57 [31 to 67] | 63 [39 to 72] | 60 [23 to 76] | 60 [23 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 6 | 24
  Male | 5 | 7 | 9 | 21
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 15 | 45

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients Who Had a 50% or Greater Wound Size Volume Reduction After 4 Weeks of Treatment With the Next Science Wound Gel, as Compared to Wounds Treated With Standard of Care
Time Frame: Percentage after 4 weeks
Measure: Number; unit: percentage of participants
Arm/Group | NXTSC | NXTSC Plus SOC | Standard of Care
Number analyzed (Participants) | 15 | 15 | 15
percentage of participants | 62 | 72 | 47

ADVERSE EVENTS:
Arm/Group | NXTSC | NXTSC Plus SOC | Standard of Care
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes